CLINICAL TRIAL: NCT03933696
Title: Light, Metabolic Syndrome and Alzheimer's Disease: A Non-Pharmocological Approach
Brief Title: Light, Metabolic Syndrome and Alzheimer's Disease - Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Population Health Science and Policy, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 17-2685-0002
Record Dates: First submitted 2019-04-25; First posted 2019-05-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Type2 Diabetes
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive the active or placebo lighting condition
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Lighting Intervention (Active Comparator): The TLI will provide high circadian stimulation during the day produced by light sources that provide moderate light levels of spectra that are tuned to the sensitivity of the circadian system. Combining spectrum and light level, TLI will allow us to: (a) use a light source that will stimulate the circadian system, and (b) provide the participants with options as to how the light treatment will be delivered. The investigators will deliver at least 300-400 lux at the eye of the bluish-white light during the day (CS of 0.4 or greater).
  The lighting intervention will be in place for 24 weeks
  Interventions: Device: Tailored Lighting Intervention
- Placebo Lighting Intervention (Placebo Comparator): The placebo condition light source will be a warm yellow - white (2700 - 3000 K) source providing 50 -100 lux at the eye. The lighting intervention will be in place for 24 weeks.
  Interventions: Device: Tailored Lighting Intervention

INTERVENTIONS:
Device: Tailored Lighting Intervention — Lighting Intervention either Active or Placebo

SUMMARY:
To test the long term effect of a light treatment on cognition, sleep and metabolism in patients with Mild cognitive impairment (MCI) or mild Alzheimer's disease or related dementia (ADRD).

DETAILED DESCRIPTION:
Test if a tailored light intervention (TLI) that promotes entrainment can improve sleep disturbances, inflammation, insulin sensitivity (Si) and glucose disposal (Sg) and cognition in patients with MCI and mild ADRD and sleep disturbances. Using a single-arm, between-subjects, placebo-controlled study the investigators will investigate if long-term (6-month) exposure to TLI improves glucose homeostasis and insulin sensitivity in patients with MCI and mild AD who suffer from sleep disturbance and are living at home. Participants will be recruited from the Mount Sinai AD research center (ADRC) and randomized to receive the TLI (or comparison control treatment) at home. The investigators hypothesize that, compared to the comparison light, a TLI will increase entrainment, improve sleep, reduce depression, reduce inflammation, improve metabolic control, increase insulin sensitivity, and reduce susceptibility to T2DM and metabolic disease during and after the completion of the 6-month intervention.

ELIGIBILITY:
Inclusion Criteria:

* Mild cognitive impairment
* Mild Alzheimer's Disease
* Sleep Disturbance
* Live at home

Exclusion Criteria:

* Blindness
* insulin-dependent diabetes patients
* macular degeneration
* severe sleep apnea

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Metabolic control | Done at Baseline, week 13 and 25
  Changes in glucose homeostasis and insulin sensitivity will be measured using the Frequently Sampled Intravenous Glucose Tolerance Test (FSIVGTT).

SECONDARY OUTCOMES:
Sleep disturbance using actigraphy | Done at Baseline, week 13, 25 and 48
  Actigraphs will be worn for 7 days during assessment weeks to measure sleep
Light measurements | Done at Baseline, week 13, 25 and 48
  Light measurements will be collected using the Daysimeter for 7 days.
Melatonin Levels | One morning during Baseline, week 13, 25 and 48
  First morning urine will be collected and assayed for melatonin levels
Sleep disturbance | Done at Baseline, week 13, 25 and 48
  Change in sleep disturbance will be assessed using the Pittsburgh Sleep Quality Index. The sum of the 7 component scores yields a single global score. A person with a global score above 5 is considered to have sleep disturbances. A higher score indicates worsening sleep disturbance.
Depression | Done at Baseline, week 13, 25 and 48
  A change in depression will be assessed using the Cornell Scale for Depression in Dementia. A score of nine or more points indicates depression.
Cognition | Done at Baseline, week 13, 25 and 48
  Changes in cognition will be assessed by use of the Alzheimer's Disease Assessment Scale- Cognitive Sub scale (ADAS-Cog). Scores range from 0 to 70 and a higher score signifies a greater degree of cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana G Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Rutgers University, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No